CLINICAL TRIAL: NCT06246357
Title: Phase 2 Study Evaluating the Functional Status of the Adrenal Glands With [68Ga]Ga-PentixaFor in Hyperaldosteronism and Hypercortisolism
Brief Title: Evaluating the Functional Status of the Adrenal Glands With [68Ga]Ga-PentixaFor in Hyperaldosteronism and Hypercortisolism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10001600; 001600-C
Record Dates: First submitted 2024-02-06; First posted 2024-02-07 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12-05

CONDITIONS: Hyperaldosteronism; Hypercortisolism; Cushing s Syndrome
Keywords: Adenomas; PET Imaging
MeSH Terms: conditions — Hyperaldosteronism; Cushing Syndrome; Adenoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/[68Ga]Ga-PentixaFor PET/CT or PET/MR (Experimental): Participants will undergo [68Ga]Ga-PentixaFor PET/CT or PET/MR
  Interventions: Drug: [68Ga]Ga-PentixaFor

INTERVENTIONS:
Drug: [68Ga]Ga-PentixaFor — [68Ga]Ga-PentixaFor will be injected intravenously approximately 60 minutes prior to scanning at a dose of 150 +/- 50 MBq (4 mCi +/- 1.4).

SUMMARY:
Background:

The adrenal glands are 2 small organs that sit on top of each kidney. They release hormones; these are chemicals that control how the body works. Tumors on or outside the adrenal glands are called functional if they release hormones; they are called nonfunctional if they do not. Doctors who treat adrenal tumors need to know which type a person has. Researchers want to find better ways to learn whether an adrenal tumor is functional.

Objective:

To see if a new radioactive tracer ([68Ga]Ga-PentixaFor) can make it easier to identify functional adrenal tumors with positron emission tomography (PET) scans.

Eligibility:

People aged 18 years and older with 1 or more adrenal tumors. They must have increased levels of the hormones aldosterone or cortisol. They must also be enrolled in at least 1 other related NIH study (protocols 19-DK-0066, 18-CH-0031, or 09-C-0242).

Design:

Participants will be screened. They may have imaging scans. Their ability to perform normal activities will be reviewed.

Participants will have one PET scan with the study tracer.

The tracer will be given through a tube attached to a needle inserted into a vein. Participants will receive the tracer 1 hour before the scan. They will lie still on a bed while a machine captures images of the inside of their body. The scan will take 45 to 90 minutes.

Participants heart rate, blood pressure, and rate of breathing will be checked before, during, and after the scan.

Participants will have a follow-up visit 3 days after their scan. This visit can be by phone, email, or in person.

DETAILED DESCRIPTION:
Background:

* [68Ga]Ga-PentixaFor is a PET agent targeting the C-X-C chemokine receptor type 4 (CXCR4) with promising applications in oncology, cardiology, and infectious disease.
* CXCR4 has also been noted to show high expression in many aldosterone-producing adenomas (APA) and some cortisol-producing adenomas (CPA) but not usually in nonfunctioning adenomas.
* [68Ga]Ga-PentixaFor may be useful in the evaluation of adrenal adenomas in the setting of Conn's or Cushing's syndrome. Localizing functional adenomas is important for managing treatment options but current imaging modalities are either too invasive or insufficiently able to differentiate adrenal conditions.

Objective:

-To estimate the percent concordance of [68Ga]Ga-PentixaFor imaging with clinical diagnosis in identifying functional adrenal or extra-adrenal adenomas in hyperaldosteronism and hypercortisolism

Eligibility:

* Must have any of the following:

  * one or more adrenal masses on CT and/or MRI and biochemical evidence of excess aldosterone or
  * ACTH-independent hypercortisolism with or without adrenal masses on CT and/or MRI or
  * history of ACTH-dependent hypercortisolism (with or without adrenal enlargement)
* Age >= 18 years
* ECOG performance status <= 2

Design:

* This is a Phase II, single site study where participants from three cohorts are enrolled into one arm according to their probable disease: primary aldosteronism (Cohort 1), ACTHindependent Cushing's syndrome (Cohort 2), or ACTH-dependent Cushing's syndrome (Cohort 3).
* All participants will undergo a [68Ga]Ga-PentixaFor PET/CT or [68Ga]Ga-PentixaFor PET/MR.
* A safety visit will be performed 3 days following the [68Ga]Ga-PentixaFor imaging.
* Participants will remain on-study for up to 1 year to allow the collection of samples for correlative analysis from the parent protocol (adrenal venous sampling, imaging assessments, laboratory evaluations, and/or tissue samples).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have any of the following:

  * one or more adrenal masses on CT and/or MRI and biochemical evidence of excess aldosterone

OR

--ACTH-independent hypercortisolism, with or without adrenal masses on CT and/or MRI

OR

* history of ACTH-dependent hypercortisolism (with or without adrenal enlargement)
* Co-enrollment in 19-DK-0066, 09-C-0242, 18-CH-0031 or a similar NIH trial.
* Age >=18 years.
* ECOG performance status <= 2.
* Women of child-bearing potential (WOCBP) and men must agree to use an effective contraception (barrier, hormonal, intrauterine device [IUD], surgical sterilization, abstinence) for two weeks prior to [68Ga]Ga-PentixaFor scan and for one week after the [68Ga]Ga-PentixaFor scan.

  * Breastfeeding should be discontinued for one week after the [68Ga]Ga-PentixaFor scan.
  * Men must agree not to donate sperm for one week after the [68Ga]Ga-PentixaFor scan.
* Participants must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Positive beta-human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test performed in females of childbearing potential at screening.
* Uncontrolled intercurrent illness or social situations based on the review of medical history that would limit compliance with study requirements.
* Contraindications to having an MRI and CT.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the percent concordance of [68Ga]Ga-PentixaFor imaging with clinical diagnosis in identifying functional adrenal or extra-adrenal adenomas in hyperaldosteronism and hypercortisolism | Screening
  The percent concordance between [68Ga]Ga-PentixaFor and clinical diagnosis will be estimated within each Cohort, along with 90% Clopper-Pearson confidence intervals.

SECONDARY OUTCOMES:
Compare [68Ga]Ga-PentixaFor uptake to C-X-C chemokine receptor type 4 (CXCR4) expression in resected tissue (when obtained on parent protocol) | Within 1 year following [68Ga]Ga-PentixaFor imaging
  The Spearman rank correlation coefficient between [68Ga]Ga-PentixaFor PET parameters (SUVmax, SUVmean, TLU, TV) and CXCR4 expression as measured via immunohistochemistry will be estimated within each Cohort.
Evaluate threshold values of [68Ga]Ga-PentixaFor uptake for determining adrenal mass hyperfunction | Within 1 year following [68Ga]Ga-PentixaFor imaging
  Receiver operating characteristic (ROC) curves of [68Ga]Ga-PentixaFor SUVmax in detecting adrenal mass hyperfunction will be constructed. The cutoff associated with the highest Youden index (sensitivity plus specificity) will be selected as the optimal threshold.
Estimate the safety of [68Ga]Ga-PentixaFor | Day of [68Ga]Ga-PentixaFor administration until end of study participation
  Safety will be evaluated by determining the frequency of adverse events among participants and reporting the results, by maximum grade of event and type of toxicity noted.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Liza Lindenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001600-C.html